CLINICAL TRIAL: NCT05261295
Title: Comparison of PEEP Applying in Terms of Perioperative Oxygenation and Postoperative Pulmonary Complications in the Use of Classical LMA and I-gel in Urological Surgery Procedures in Lithotomy Position
Brief Title: Comparison of PEEP Effect on Perioperative Oxygenation and Postoperative Pulmonary Complications in Lithotomy Position
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, canan ün, principal investigator, Ankara City Hospital Bilkent
Other Study IDs: E1-21-2260
Record Dates: First submitted 2022-02-11; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Positive End Expiratory Pressure; Lung Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Classical LMA: Patients who received general anesthesia with classical LMA
  Interventions: Diagnostic Test: PEEP; Diagnostic Test: ZEEP
- i-Gel: Patients who received general anesthesia with i-Gel
  Interventions: Diagnostic Test: PEEP; Diagnostic Test: ZEEP

INTERVENTIONS:
Diagnostic Test: PEEP — PEEP of 7 cmH2O will be applied 5 minutes after classical LMA or i-gel insertion.
Diagnostic Test: ZEEP — PEEP of 0 cmH2O will be applied 5 minutes after classical LMA or i-gel insertion.

SUMMARY:
The main purpose of the study is to compare the effectiveness of PEEP application in terms of perioperative oxygenation level in the use of classical LMA and i-gel, which is often preferred. The secondary aim is to compare parameters such as gastric insufflation and the rate of postoperative pulmonary complication development in the case of PEEP with two supraglottic airway devices.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Patients who will undergo transurethral resection of the bladder and prostate taken in the lithotomy position, ureter and kidney stone operations with ureteroscopy

Exclusion Criteria:

* Heart failure (ejection fraction < 40%),
* unstable hemodynamic conditions
* Having neck or upper respiratory tract pathology,
* have an increased risk of aspiration (gastroesophageal reflux disease, full stomach, acidity),
* obesity (body mass index≥30 kg m-2)
* Patients with poor tooth structure will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo transurethral resection of the bladder and prostate taken in the lithotomy position, ureter and kidney stone operations with ureteroscopy
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
LUS score preop | Baseline
  Loss of ventilation will be evaluated by calculating the LUS score. Each region will be scored according to the LUS model as follows: Presence of lung deviation with lines or less than two isolated B-lines is scored as 0; 1 point in the presence of more than one well-defined B line; presence of more than one combined B line, 2 points; and when a tissue pattern characterized by dynamic air bronchograms (lung consolidation) is presented, the score is 3. The worst ultrasound pattern observed in each region will be recorded and used to calculate the sum of the scores.
LUS score postoperative | postoperative 1.hour
  Loss of ventilation will be evaluated by calculating the LUS score. Each region will be scored according to the LUS model as follows: Presence of lung deviation with lines or less than two isolated B-lines is scored as 0; 1 point in the presence of more than one well-defined B line; presence of more than one combined B line, 2 points; and when a tissue pattern characterized by dynamic air bronchograms (lung consolidation) is presented, the score is 3. The worst ultrasound pattern observed in each region will be recorded and used to calculate the sum of the scores.

CONTACTS AND LOCATIONS:
Overall Officials: canan ün, MD, Principal Investigator — ankara ch bilkent

IPD SHARING:
Plan to Share IPD: Undecided